CLINICAL TRIAL: NCT01901809
Title: Randomized Evaluation of Heart Failure With Preserved Ejection Fraction (HFpEF) Patients With Acute Heart Failure and Dopamine (ROPA-DOP) Trial
Brief Title: Diuretics and Dopamine in Heart Failure With Preserved Ejection Fraction
Acronym: ROPA-DOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NA 00083629
Record Dates: First submitted 2013-05-15; First posted 2013-07-17 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure, Diastolic
Keywords: Heart failure, diastolic; HFpEF; Diuretics; Dopamine
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Furosemide; Dopamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bolus furosemide and no dopamine (Active Comparator): If the patient is not on a prior diuretic dose, a standard dose of furosemide 40mg IV every 12 hrs, with total dose of 80 mg IV over 24 hrs will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose every 12 hrs. (i.e if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose will be furosemide 80mg IV twice daily).
  Interventions: Drug: Furosemide
- Continuous infusion furosemide and no dopamine (Active Comparator): If the patient is not on a prior diuretic dose, a standard dose of furosemide 80mg IV over 24 hrs, will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose continuously over 24 hrs. . (i.e. if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose would be furosemide 160mg IV to be administered continuously over 24 hrs).
  Interventions: Drug: Furosemide
- Bolus furosemide plus dopamine (Active Comparator): Intermittent furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min
  Interventions: Drug: Furosemide; Drug: Dopamine
- Continuous furosemide plus dopamine (Active Comparator): Continuous furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min
  Interventions: Drug: Furosemide; Drug: Dopamine

INTERVENTIONS:
Drug: Furosemide
Drug: Dopamine
  Arms: Bolus furosemide plus dopamine; Continuous furosemide plus dopamine

SUMMARY:
Heart Failure with preserved Ejection Fraction (HFPEF) accounts for 40-50% of all heart failure patients with a frequency of hospital admissions for acute decompensation and short and long term mortality similar to patients with heart failure with reduced ejection fraction (HFREF). Patients with HFPEF are often preload dependent and despite admission to the hospital for acute decompensated heart failure (ADHF), are typically difficult to diurese due to the development of acute kidney injury. No studies have been performed evaluating treatment strategies for these patients. The investigators hypothesize that changing the method of diuresis and/or the addition of low-dose dopamine for the treatment of ADHF in patients with HFPEF will reduce renal injury, resulting in a shorter length of stay, and decrease hospital readmissions over the ensuing year. This trial will randomize patients to either bolus or continuous infusion furosemide and then to either dopamine or no dopamine. The primary endpoint will be renal function at 72 hours as measured by change in Glomerular Filtration Rate (GFR). Secondary endpoints for readmission, functional capacity, quality of life, and amount of diuresis will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Johns Hopkins Hospital for acute decompensated heart failure.
* Patient ≥18 years of age
* Estimated GFR of > 15 milliliters/min/1.73m2 determined by the Modification of Diet in Renal Disease (MDRD) equation
* Willingness to provide informed consent
* Known ejection fraction by noninvasive testing of > 50% within 12 months of admission to the hospital with no interval myocardial infarction since inclusion transthoracic echo, by history, or by ECG.
* Negative pregnancy test in a female of child bearing potential
* Willingness of primary attending physician for patient to participate.

Exclusion Criteria:

* Systolic BP <90 mmHg on admission
* Hemoglobin (Hgb) < 8 g/dl
* Known allergy or intolerance to furosemide or low dose dopamine.
* Hemodynamically significant arrhythmias including ventricular tachycardia or defibrillator shock within 4 weeks
* Acute coronary syndrome within 4 weeks
* Cardiac diagnoses in addition to or other than HFpEF:

  i. Active myocarditis ii. Hypertrophic obstructive cardiomyopathy iii. Severe valvular disease iv. Restrictive or constrictive cardiomyopathy, including known amyloidosis, sarcoidosis, hemachromatosis v. Complex congenital heart disease vi. Constrictive pericarditis vii. Severe pulmonary hypertension (RVSP ≥ 60), not secondary to HFpEF
* Non-cardiac pulmonary edema
* Clinical evidence of digoxin toxicity
* Received IV vasoactive treatment or ultra-filtration therapy for heart failure since initial presentation
* Anticipated need for IV vasoactive treatment or ultra-filtration for heart failure during this hospitalization
* History of temporary or permanent renal replacement therapy or ultrafiltration
* History of renal artery stenosis > 50%
* Need for mechanical hemodynamic support
* Sepsis
* Terminal illness (other than HF) with expected survival of less than 1 year
* Previous adverse reaction to the study drugs
* Use of IV iodinated contrast material/dye in last 72 hours or planned during hospitalization
* Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
* Inability to comply with planned study procedures
* Pregnancy or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Kavita, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Rasoul D, Zhang J, Farnell E, Tsangarides AA, Chong SC, Fernando R, Zhou C, Ihsan M, Ahmed S, Lwin TS, Bateman J, Hill RA, Lip GY, Sankaranarayanan R. Continuous infusion versus bolus injection of loop diuretics for acute heart failure. Cochrane Database Syst Rev. 2024 May 22;5(5):CD014811. doi: 10.1002/14651858.CD014811.pub2. PMID 38775253
- [Derived] Sharma K, Vaishnav J, Kalathiya R, Hu JR, Miller J, Shah N, Hill T, Sharp M, Tsao A, Alexander KM, Gupta R, Montemayor K, Kovell L, Chasler JE, Lee YJ, Fine DM, Kass DA, Weiss RG, Thiemann DR, Ndumele CE, Schulman SP, Russell SD; Osler Medical Housestaff. Randomized Evaluation of Heart Failure With Preserved Ejection Fraction Patients With Acute Heart Failure and Dopamine: The ROPA-DOP Trial. JACC Heart Fail. 2018 Oct;6(10):859-870. doi: 10.1016/j.jchf.2018.04.008. Epub 2018 Aug 8. PMID 30098962

RESULTS

PARTICIPANT FLOW:
Groups:
- Bolus Furosemide: If the patient is not on a prior diuretic dose, a standard dose of furosemide 40mg IV every 12 hrs, with total dose of 80 mg IV over 24 hrs will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose every 12 hrs. (i.e if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose will be furosemide 80mg IV twice daily).
  Furosemide
- Continuous Infusion Furosemide: If the patient is not on a prior diuretic dose, a standard dose of furosemide 80mg IV over 24 hrs, will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose continuously over 24 hrs. . (i.e. if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose would be furosemide 160mg IV to be administered continuously over 24 hrs).
  Furosemide
- Bolus Furosemide Plus Dopamine: Intermittent furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min administered as an infusion.
  Furosemide
  Dopamine
- Continuous Furosemide Plus Dopamine: Continuous furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min administered as an infusion.
  Furosemide
  Dopamine
Period: Overall Study
Arm/Group | Bolus Furosemide | Continuous Infusion Furosemide | Bolus Furosemide Plus Dopamine | Continuous Furosemide Plus Dopamine
Started | 19 | 23 | 24 | 24
Completed | 19 | 23 | 21 | 22
Not Completed | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bolus Furosemide | Continuous Infusion Furosemide | Bolus Furosemide Plus Dopamine | Continuous Furosemide Plus Dopamine | Total
Number analyzed (Participants) | 19 | 23 | 24 | 24 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 12 | 11 | 42
  >=65 years | 10 | 13 | 12 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (13) | 63 (10) | 66 (15) | 67 (13) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 17 | 15 | 61
  Male | 2 | 11 | 7 | 9 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 12 | 14 | 15 | 15 | 56
  White | 6 | 9 | 9 | 9 | 33
  Other | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum Creatinine at 72 Hours.
Description: Percent change in serum creatinine from randomization to 72 hrs from treatment protocol initiation.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: percent change in serum creatinine
Groups:
- Bolus Furosemide and no Dopamine: If the patient is not on a prior diuretic dose, a standard dose of furosemide 40mg IV every 12 hrs, with total dose of 80 mg IV over 24 hrs will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose every 12 hrs. (i.e if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose will be furosemide 80mg IV twice daily).
  Furosemide
- Continuous Infusion Furosemide and no Dopamine: If the patient is not on a prior diuretic dose, a standard dose of furosemide 80mg IV over 24 hrs, will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose continuously over 24 hrs. . (i.e. if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose would be furosemide 160mg IV to be administered continuously over 24 hrs).
  Furosemide
- Bolus Furosemide Plus Dopamine: Intermittent furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min
  Furosemide
  Dopamine
- Continuous Furosemide Plus Dopamine: Continuous furosemide diuretic therapy as outlined with the addition of dopamine at 3 µg/kg/min
  Furosemide
  Dopamine
Arm/Group | Bolus Furosemide and no Dopamine | Continuous Infusion Furosemide and no Dopamine | Bolus Furosemide Plus Dopamine | Continuous Furosemide Plus Dopamine
Number analyzed (Participants) | 19 | 23 | 24 | 24
percent change in serum creatinine | 4 (22) | 11 (21) | 5 (17) | 20 (28)

2. Primary Outcome: Percent Change in Serum Creatinine at 72 Hours - Continuous vs Intermittent Diuretic
Description: Percent change in serum creatinine from randomization to 72 hrs from treatment protocol initiation by diuretic strategy
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: percent change in serum creatinine
Groups:
- Bolus Furosemide: If the patient is not on a prior diuretic dose, a standard dose of furosemide 40mg IV every 12 hrs, with total dose of 80 mg IV over 24 hrs will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose every 12 hrs. (i.e if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose will be furosemide 80mg IV twice daily).
- Continuous Infusion Furosemide: If the patient is not on a prior diuretic dose, a standard dose of furosemide 80mg IV over 24 hrs, will be initiated.
  If the patient is already on a prescribed diuretic dose, their outpatient dose will be doubled and administered as the equivalent IV dose continuously over 24 hrs. . (i.e. if the prescribed dose is furosemide 80mg by mouth twice daily, the inpatient treatment dose would be furosemide 160mg IV to be administered continuously over 24 hrs).
Arm/Group | Bolus Furosemide | Continuous Infusion Furosemide
Number analyzed (Participants) | 43 | 47
percent change in serum creatinine | 4.6 [-1.1 to 10.4] | 16 [8.5 to 23.4]
Statistical Analysis 1: Comparison: Bolus Furosemide vs Continuous Infusion Furosemide; Test type: Superiority; p = 0.018, t-test, 2 sided; Mean Difference (Net) = 11.4, 95% CI 2-sided [2.0 to 20.8], Standard Error of Mean 4.7

3. Primary Outcome: Percent Change in Serum Creatinine at 72 Hours - Dopamine vs No Dopamine
Description: Percent change in serum creatinine from randomization to 72 hrs from treatment protocol initiation by dopamine strategy
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: percent change in serum creatinine
Groups:
- Dopamine: Diuretic therapy plus addition of dopamine at 3 µg/kg/min administered as an infusion.
- No Dopamine: Diuretic therapy only
Arm/Group | Dopamine | No Dopamine
Number analyzed (Participants) | 48 | 42
percent change in serum creatinine | 8.0 [1.4 to 14.6] | 12.8 [5.7 to 20.0]
Statistical Analysis 1: Comparison: Dopamine vs No Dopamine; Test type: Superiority; p = 0.33, t-test, 2 sided; Mean Difference (Net) = -4.8, 95% CI 2-sided [-14.4 to 4.9], Standard Error of Mean 4.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bolus Furosemide | Continuous Infusion Furosemide | Bolus Furosemide Plus Dopamine | Continuous Furosemide Plus Dopamine
All-Cause Mortality (participants affected / at risk) | 5/19 | 3/22 | 4/23 | 3/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22 | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. The investigator team was blinded to study assignment; however, the patient and treating physicians were un-blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT01901809/Prot_SAP_000.pdf